CLINICAL TRIAL: NCT02847663
Title: The Effect of Whole Body Cryotherapy on Recovery and Performance: a Randomized Controlled Trial
Acronym: Cryotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences and Arts of Southern Switzerland (Other)
Collaborators: THIM - die internationale Hochschule für Physiotherapie (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Ron Clijsen, PhD., University of Applied Sciences and Arts of Southern Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PB_2016-01125
Record Dates: First submitted 2016-06-15; First posted 2016-07-28 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Cold
Keywords: Cold; recovery
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole-body cryotherapy (Experimental): The effects of whole-body cryotherapy (-135°C for 2 minutes) are investigated after a muscle damage protocol.
  Interventions: Device: Kryosauna Space Cabin
- Cold-water immersion (Other): The effects of cold-water immersion (10°C for 15 minutes) are investigated after a muscle damage protocol.
  Interventions: Other: cold water tub

INTERVENTIONS:
Device: Kryosauna Space Cabin — The whole body cryotherapy device is able to generatue temperatures up to -195°C for 3 minutes. In this study, we generate temperatures of -135°C for 2 minutes as proposed in the manual. The participant will enter the cabin in cold-resistant shoes and will remain in standing position during the whole procedure. The cold temperature is generated by vaporization of liquid nitrogen.
  Other Names: Cryomed s.r.o.
  Arms: Whole-body cryotherapy
Other: cold water tub — The tub will be filled with cold water up to the sternal level of the participants. Adding ice will ensure a constant temperature. The participant will sit inside the tub during the whole procedure.
  Arms: Cold-water immersion

SUMMARY:
This study investigates the effects of whole-body cryotherapy vs. cold-water immersion after a muscle damage protocol.

DETAILED DESCRIPTION:
In this study the effects of a single- or multiple whole body cryotherapy (-135°C for max. 2 minutes) vs. cold water immersion (10°C for 15 min) and a passive control group (20 min supine position) are compared. These effects are examined after a muscle damage protocol of the frontal thighs (3 x 30 jumps). The objective recovery parameters are vertical jump, maximum voluntary contraction of the anterior thigh muscle, heart rate, blood pressure, skin-core body temperature and the oxygen saturation of the thigh muscles. Subjective recovery parameters are the local muscle soreness details and the general exhaustion details. The parameters are directly and 24, 48 and measured 72 hours after exposure. The aim is to elicit the effects of whole body cooling to make recommendations to. The current scientific knowledge situation calls for further studies to whole body cooling.

ELIGIBILITY:
Inclusion Criteria:

Only healthy young subjects 18-35 years no musculoskeletal surgery in trunk and lower extremities injury history in trunk and lower extremity for more than one year subjects taking anticonceptive medication are allowed to participate

Exclusion Criteria:

Actual injuries or injuries for less than one year in trunk and /or lower extremities injury history in trunk and lower extremity for more than one year with complaints anxiety of cooling subjects on medication pace maker cardiovascular disease pregnancy skeletal problems appendectomy for less than two years Morbus Raynaud syndrome

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Vertical Jump | 72 hours
  Vertical Jump will be assessed in cm with the Just Jump Plate
Maximum voluntary contraction | 72 hours
  Maximum voluntary contraction will be assessed in kg on a custom made ergometer chair (COR 1)
Delayed onset of muscle soreness | 72 hours
  DOMS will be assessed using a visual analog scale (0-10 cm)
Ratings of perceived exertion | 72 hours
  RPE will be assessed using a BORG scale (6-20)
Skin temperature | 60 minutes
  Skin temperature of the neck, right scapula, right dorsal hand, right frontal thigh, right shin are assessed in °C using thermocouples (iButtons)
Core temperature | 60 minutes
  Core temperature will be assessed in °C via the ear
Cardiovascular measurements | 60 min
  Heart rate will be measured in beats per minute and bloop pressure will be measured in mm/Hg using an blood pressure monitor
Oxygenation of the right thigh muscle | 60 min
  Oxygenation of the right thigh muscle will be assessed in % using a near infrared spectometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ronaldus Clijsen, PhD, Principal Investigator — Fachhochschule Südschweiz
Locations (1):
- Fachhochschule Südschweiz, Landquart, Switzerland

IPD SHARING:
Plan to Share IPD: No